CLINICAL TRIAL: NCT03064594
Title: Comparison of Laparoscopic Cornuostomy and Wedge Resection for Interstitial Pregnancy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 105143-E
Record Dates: First submitted 2017-02-09; First posted 2017-02-27 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cornual Pregnancy
MeSH Terms: conditions — Pregnancy, Cornual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cornuostomy: cornuostomy
  Interventions: Procedure: Cornual pregnancy
- wedge resection: wedge resection

INTERVENTIONS:
Procedure: Cornual pregnancy — we will get the information of operative time, blood loss and postoperative pregnancy and delivery rate.
  Groups: cornuostomy

SUMMARY:
This retrospective study is to find out the best way to treat patient with cornual pregnancy in the aspect of further pregnancy outcome.

DETAILED DESCRIPTION:
To find out the best way to treat patient with cornual pregnancy in the aspect of further pregnancy outcome, the investigators compared the outcomes of laparoscopic wedge resection (LWR) and laparoscopic cornuostomy (LC) by the retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* All women with cornual pregnancy who were admitted to the Department of Obstetrics and Gynecology of the Far Eastern Memorial Hospital for laparoscopic surgeries between January 2008 and June 2016 were enrolled

Exclusion Criteria:

* The person who was pregnant at the time of the operation
* After receiving IVF course of treatment
* Patients with uterine horns undergoing open surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the cases with cornual pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 9 years
  Comparison of pregnancy rates between the cornuostomy and wedge resection groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, New Taipei City, Banqiao, Taiwan